CLINICAL TRIAL: NCT04199676
Title: Immediate Postpartum Glucose Tolerance Testing Among Gestational Diabetics: A Comparison to the Gold Standard
Brief Title: Immediate Postpartum Glucose Tolerance Testing
Status: Recruiting | Type: Observational
Sponsor: MemorialCare Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 925-19
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood specimens will be obtained as part of the glucose tolerance testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: 75g glucose tolerance test to be administered during postpartum hospitalization
  Interventions: Diagnostic Test: Glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Glucose tolerance test — Oral administration of a 75g glucose tolerance test during the postpartum hospitalization

SUMMARY:
The objective of this study is to compare the accuracy of a 2hr glucose tolerance test administered during the postpartum hospitalization with the standard of care glucose tolerance testing (administered at 6 weeks postpartum). The primary hypothesis is that the glucose tolerance test administered in the postpartum period will be accurate and will improve compliance with postpartum testing for gestational diabetics.

DETAILED DESCRIPTION:
Gestational diabetes affects approximately 5-10% of pregnancies and its prevalence continues to increase as rates of obesity and metabolic disease increase in reproductive age women. Women diagnosed with gestational diabetes carry an increased risk of developing type 2 diabetes later in life, even if their glucose tolerance initially normalizes following delivery.

The gold standard assessment of glucose tolerance postpartum is a two hour glucose tolerance test (GTT) that is completed between six and twelve weeks' postpartum. Unfortunately, the compliance rate with this test is low, ranging from 30 - 50% by most reports. As a result, a large number of women with glucose intolerance are missed due to noncompliance with postpartum testing, thereby forfeiting the opportunity for diagnosis, treatment and prevention of longterm health consequences. The postpartum hospital stay provides a unique opportunity to increase compliance with glucose tolerance testing due to an increased rate of patient capture. However, it is unknown if administration of a glucose tolerance test in the immediate postpartum period would adequately identify women with persistent glucose intolerance.

The current study aims to provide data towards the accuracy of an immediate postpartum GTT in a population of women with gestational diabetes and provide follow-up data on women with abnormal testing.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or recently postpartum (postpartum day 0 or 1)
* ≥ 18 years of age
* Gestational age ≥34 weeks
* A1 or A2 gestational diabetes

Exclusion Criteria:

* Medical exclusion from completing glucose tolerance testing
* Steroid administration within 10 days prior to enrollment
* Chronic steroid use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All individual diagnosed with gestational diabetes will be approached following admission to labor and delivery and invited to participate.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of immediate glucose tolerance testing | 6-12 weeks postpartum
  Diagnostic accuracy between immediate postpartum glucose tolerance testing and gold standard testing

SECONDARY OUTCOMES:
Compliance with standard glucose tolerance testing | 12 weeks postpartum
  Percentage of the cohort that comply with glucose tolerance testing at their postpartum visit
Transition to primary care | 12 weeks postpartum
  Percentage of cohort that are appropriately referred to ongoing primary care

CONTACTS AND LOCATIONS:
Overall Officials: Alice Sherman-Brown, MD, Principal Investigator — Magella Medical Group
Locations (1):
- Long Beach Memorial Medical Center/Miller Children's and Women's Hospital, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: Undecided